CLINICAL TRIAL: NCT05190354
Title: Post Market Clinical Protocol - Xtremity Polymer Prosthetic Socket System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Creations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP-0001
Record Dates: First submitted 2021-12-06; First posted 2022-01-13 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Amputation; Prosthesis User
Keywords: transtibial; amputation; prosthesis; below knee

STUDY DESIGN:
Intervention Model Description: Subjects with transtibial unilateral or bilateral amputation who have experience using carbon fiber or high temperature thermoplastic prosthetic socket and are at least 6-months post-amputation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Xtremity Prosthesis (Experimental): Xtremity Prosthesis fitting
  Interventions: Device: Xtremity Polymer Prosthetic Socket

INTERVENTIONS:
Device: Xtremity Polymer Prosthetic Socket — Subjects with transtibial unilateral or bilateral amputation who have experience using a standard carbon fiber or high temperature thermoplastic prosthetic socket will be evaluated and fitted with a below knee prosthesis socket

SUMMARY:
Single-arm, prospective multi-center study assessing user preference of the Xtremity prosthetic socket in below the knee amputation prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 19 years old
* Unilateral or bilateral transtibial amputation
* Subject has been informed of the nature of the study, agrees to participate and comply with all follow-up visits and has signed the consent form.
* Currently using a standard carbon fiber or high temperature thermoplastic prosthetic socket.
* Residual limb is between 26-34 cm circumference with a liner (when measured 4cm proximal to distal end)
* Subject is eligible for standard carbon fiber or high temperature thermoplastic prosthetic socket if necessary.
* Must be able to ambulate at least 100 yards with or without an assistive device.
* Must be able to don and doff a prosthesis independently.
* Estimated life expectancy > 1 year

Exclusion Criteria:

* Amputation < 6 months prior to enrollment
* Residual limb less than (<) 26cm and greater than (>) 34cm circumference at the distal end.
* Body weight greater than (>) 275lbs.
* Syme's amputations or total limb length over 30cm
* Some bulbous or irregular limb shapes
* Build height and circumference limitations
* Wounds or skin issues that preclude normal fit
* Unusual alignment of the socket or foot
* Alignment outside the capability of the Xtremity System.
* Planned for any major surgery within 6 months of enrollment.
* Subject is pregnant or breastfeeding
* Subject is incarcerated.
* Subject anticipates that the socket will frequently be subject to temperatures greater than 110 degrees F while in their possession.
* Subject anticipates that the socket will frequently be subject to direct sunlight
* Limb circumference at the mid-patella tendon exceeds the maximum circumference (see sizing chart in the instructions for use)
* Subject is participating in another research study of a device, medication, which could, in the opinion of the investigator, affect the results of this study.
* Subject has other medical, social or psychological problems that in the opinion of the investigator would preclude them from receiving this treatment and the procedures and or participating in evaluations pre and post-treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
User Preference of the Xtremity Socket - Achievement of durability | 21 days
  Device success defined as rate of achieving durability
User Preference of the Xtremity Socket - Socket Comfort Score | 21 Days
  Rate of device success measured by Socket Comfort Score
User Preference of the Xtremity Socket - Prosthetic Evaluation Questionnaire | 21 Days
  Rate of device success measured by abbreviated Prosthetic Evaluation Questionnaire
User Preference of the Xtremity Socket - Activity | 21 Days
  Rate of device success measured by activity level ranked low activity to high activity (1-10)

SECONDARY OUTCOMES:
Benefits to prosthetist - Casting Time | 21 days
  Measured by time from casting to delivery in days
Benefits to prosthetist - Material Consumption | 21 days
  Measured by amount of material consumed
Benefits to prosthetist - Material Waste | 21 days
  Measured by amount of material wasted
Benefits to prosthetist - Resources | 21 days
  Number of resources required to use
Benefits to prosthetist - Skill | 21 days
  Level of skill set required to use ranked on a scale from very easy to very difficult (1-5)
Benefits to prosthetist - Adjustability | 21 days
  Ease of adjustability ranked from difficult to easy (1-5)
Benefits to Patient - Mobility | 21 days
  Measured by Amputee Mobility Predictor Assessment Tool
Benefits to Patient - Cosmesis | 21 days
  Measured by Cosmesis survey question ranked from very unattractive to very attractive (1-5)
Benefits to patient - Number of Visits | 21 days
  Measured as number of visits to achieve adequate fit in days
Device Safety - Composite of Device Related Adverse Events | 21 days
  Composite of device related Adverse Events (DAE) assessed throughout 21 days after prosthetic fitting. DAE is defined as a composite of all cause death, socket site skin problems that prevent wearing a prosthetic, socket site infection, and falls due to socket malfunction that result in injury.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Berke, MS, CP, FAAOP, Principal Investigator — Medical Creations
Locations (2):
- Snell Prosthetics and Orthotic Laboratory, Little Rock, Arkansas, United States
- Barber Prosthetics, Vancouver, Canada